CLINICAL TRIAL: NCT05316064
Title: The Effects of Probiotic Against Reducing Abundance of Human Papilloma Virus (HPV) in Women
Brief Title: Reducing Abundance of Human Papilloma Virus in Women by Taking Probiotic
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: funding problem
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Min-Tze LIONG, Professor, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMRR-21-1819-61300 (IIR)
Record Dates: First submitted 2022-03-17; First posted 2022-04-07 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Human Papilloma Virus Infection
Keywords: probiotics; human papilloma virus
MeSH Terms: conditions — Papillomavirus Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic 9 log CFU/day (Experimental): Intervention consists of daily oral administration of one sachet/day of probiotic for 12 weeks, where each sachet contains 9 log CFU of probiotic.
  Interventions: Biological: probiotic
- placebo (Placebo Comparator): placebo contains primarily carrier without probiotic and it is identical in taste and appearance and appear as light-yellow powder. It is also taken by the participants for 12 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Biological: probiotic — oral administration of probiotic at 9 log CFU/day for 12 weeks to reduce vaginal abundance of HPV in women compared to placebo via the use of vaginal self-swab.
  Arms: probiotic 9 log CFU/day
Other: placebo — oral administration of primarily carrier without the probiotic for 12 weeks
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of oral administration of probiotic at 9 log colony forming unit (CFU)/day to reduce vaginal abundance of HPV in women compared to placebo via the use of vaginal self-swab.

DETAILED DESCRIPTION:
Probiotics have shown an antiviral activity and several mechanisms have been demonstrated. In respiratory tract infections (RTIs), the majority of probiotics can inhibit the most important respiratory viruses by immunomodulatory mechanisms. There are over 200 different types of viruses, which cause RTIs in humans. Human rhinoviruses (HRV) are the largest group of respiratory viruses, comprising over 150 serotypes. In humans, the predominant illness caused by HRV is the acute upper RTI, also known as the common cold. The second most common viruses infecting humans are the human enteroviruses (HEV), which are associated with clinical manifestations ranging from mild respiratory symptoms to serious conditions. Influenza viruses, respiratory syncytial virus (RSV), and adenoviruses are also major causative agents of both upper and lower RTIs. In addition, many other viruses or virus groups cause RTIs, e.g., parainfluenza viruses and coronaviruses can cause a broad spectrum of respiratory diseases, ranging from mild upper RTIs to pneumonia. In recent years, with the rapid development of high-throughput molecular techniques, several new viruses associated with respiratory diseases, such as human bocavirus, human metapneumovirus, and the new coronaviruses HKU1 and NL63, have been identified as well. Recently, COVID-19 had cause huge effect worldwide. With this, to reduce the burden and severity of this pandemic, the use of probiotic in preventing of COVID-19 has been ongoing. Probiotics also had given out significant outcome in gastroenteritis infections where a study suggested that probiotics had be effective in alleviating the duration and severity of acute rotavirus gastroenteritis. Apart from this, for viruses that cause hepatitis, skin virus infections, human immunodeficiency virus (HIV), or HPV, probiotics could directly or indirectly, help reduce their symptoms or prevent infection.

Probiotics are known as a good natural non-drug, which was widely used to boost immune cells in host to fight against infection. Generally, probiotic effects are mediated through immune regulation, particularly through balance control of proinflammatory and anti-inflammatory cytokines. The immune response is initiated by innate immunity following exposure to foreign substances or tissue injury. Innate immunity exerts protective roles in host homeostasis in part by priming adaptive immune responses against persisting insults and inducing inflammation. However, the unbalanced immune response leads to severe inflammation and uncontrolled tissue damage and disease. Probiotics have been found to enhance the innate immunity and modulate pathogen-induced inflammation via toll-like receptor-regulated signaling pathways.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active women
* Age above 26 years old
* Determined as HPV positive against L1 variant
* Willing to commit throughout the experiment

Exclusion Criteria:

* On long term medication (6 months and above) for any illnesses
* Pregnant
* Uterus and/or cervix removed
* Prior HPV vaccination
* Cervical intraepithelial neoplasia

Min Age: 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2023-11-28 (Estimated); Study Completion 2023-11-28 (Estimated)

PRIMARY OUTCOMES:
Changes in vaginal abundance of HPV of women upon administration of probiotic. | 12-weeks
  Differences in vaginal HPV abundance in women upon administration of probiotic at 9 log CFU/day compared to placebo via real-time PCR quantification of the L1 capsid gene as a conserved region of the HPV genome using consensus primers PGMY09 and PGMY1.

SECONDARY OUTCOMES:
Changes in vaginal microbiota of women upon administration of probiotic. | 12-weeks
  Differences in vaginal microbiota in women upon administration of probiotic at 9 log CFU/day compared to placebo via microbiota profiling using DNA of vaginal samples amplified for bacterial 16S rRNA and analyzed for high-throughput community sequencing.
Changes in gut microbiota of women upon administration of probiotic. | 12-weeks
  Differences in gut microbiota profiles of women on probiotic and placebo via microbiota profiling using DNA of fecal samples amplified for bacterial 16S rRNA and analyzed for high-throughput community sequencing.
Changes in vaginal health of women upon administration of probiotic via the use of questionnaire. | 12-weeks
  Differences in total scores of women upon administration of probiotic at 9 log CFU/day compared to placebo via the use of vulvovaginal symptom questionnaire (VSQ) containing 21-items on a two-point scale with higher scores indicating poorer health status.
Changes in immunity of women upon administration of probiotic 9 log CFU/day as assessed via biochemical tests. | 12-weeks
  To evaluate differences in immunity of women on probiotic and placebo in terms of blood immunity profiling via measuring concentrations of immunoglobulins such as IgA, IgG and IgM, and cytokines such as interleukin (IL)-1b, IL-4, IL-10, TNF-α and IFN-γ using commercially available ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: MingTze Liong, Doctor, Study Director — School of Industrial Technology USM; Binti Sany Salina, Doctor, Principal Investigator — Institut Perubatan & Pergigian Termaju USM
Locations (1):
- Hospital Seberang Jaya, Pulau Pinang, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu P, Mageswary MU, Nisaa AA, Samsudin SB, Rusdi NIBM, Jerip ARA, Oon CE, Sany SB, Tan CS, Zhu ZH, Liong MT. Probiotic Lactiplantibacillus plantarum Probio87 Improves Gut Microbial Profiles in HPV-Positive Women: A Randomized, Placebo-Controlled and Double-Blind Study. Mol Nutr Food Res. 2025 Nov;69(22):e70247. doi: 10.1002/mnfr.70247. Epub 2025 Aug 30. PMID 40884128
- [Derived] Xu P, Mageswary U, Nisaa AA, Balasubramaniam SD, Samsudin SB, Rusdi NIBM, Jerip ARA, Oon CE, Bakar MHA, Rajendran D, Tan JJ, Roslan FF, Sreenivasan S, Balakrishnan V, Sany SB, Tan CS, Liong MT. Probiotic reduces vaginal HPV abundance, improves immunity and quality of life in HPV-positive women: a randomised, placebo-controlled and double-blind study. Benef Microbes. 2025 May 12;16(6):667-684. doi: 10.1163/18762891-bja00079. PMID 40360161